CLINICAL TRIAL: NCT04045002
Title: Development and Effectiveness of 'MyPinkMom' Educational Intervention With Anaemia in Petaling District
Brief Title: 'MyPinkMom' Educational Intervention for Pregnant Women With Anaemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Raudah Abd Rahman, Principal Investigator, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UKM PPI/111/8/JEP-2018-674
Record Dates: First submitted 2019-07-27; First posted 2019-08-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Anaemia in Pregnancy
Keywords: 'MyPinkMom' educational intervention; haemoglobin level; dietary iron intake; knowledge level; Theory of Planned Behavior construct

STUDY DESIGN:
Intervention Model Description: Intervention group receive 'MyPinkMom' educational intervention and routine antenatal care. Control group receive routine antenatal care only
Who Masked: Outcomes Assessor
Masking Description: Respondents and investigators will aware the intervention received by respondents. The data analysers who assess research outcomes will be blinded as they would not know respondents belongs to intervention or control group as each respondent will be labelled as numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group receive 'MyPinkMom' educational intervention delivered through WhatsApp application for 2 weeks and routine antenatal care.
  Interventions: Other: 'MyPinkMom' educational intervention
- Control (No Intervention): Control group receive information on anaemia in pregnancy placed at respondents' antenatal card and routine antenatal care

INTERVENTIONS:
Other: 'MyPinkMom' educational intervention — The intervention will be carried out for 2 weeks. There will be three sessions of 'MyPinkMom' that will be delivered to respondents per week. In each session, a respective 'MyPinkMom' video with audio explanation will be delivered to respondents in intervention group through WhatsApp application. It will be delivered every alternate day per week and each video will take about 3 minutes duration. Each session has its own objective and different content.
  Each of the respondent in the intervention group will be given 'MyPinkMom' diary in which they are required to document time of iron tablet intake daily as well as time of reading of 'MyPinkMom' material in each session. At the end of the intervention, a meeting with all the respondents from the intervention group will be held for question and answer session.
  Arms: Intervention

SUMMARY:
This study will use cluster randomised controlled trial design. It will be conducted at four antenatal clinics in Petaling district, Selangor, Malaysia. Two antenatal clinics will be randomised as intervention group. Other two antenatal clinics will be the control group. The investigators will recruit 60 participants from intervention and 60 participants from control group to evaluate effectiveness of 'MyPinkMom' educational intervention. Participants from intervention group will receive usual antenatal care and 'MyPinkMom' educational intervention through WhatsApp application, while those from control group receive usual antenatal care only. The outcome measurements are mean haemoglobin level, knowledge score, Theory of Planned Behaviour (TPB) construct and dietary iron intake between intervention and control group.

DETAILED DESCRIPTION:
General objective:

To assess the effectiveness of 'MyPinkMom' educational intervention in terms of knowledge on anaemia in pregnancy, Theory of Planned Behaviour (TPB) construct to adherence of daily iron tablet intake, haemoglobin level, and dietary iron intake among pregnant women with anaemia in Petaling district.

Specific objectives:

1. To determine mean knowledge score on anaemia in pregnancy, Theory of Planned Behaviour (TPB) construct on adherence to daily iron intake, haemoglobin level and dietary iron intake of respondents from intervention and control group at baseline.
2. To compare knowledge on anaemia in pregnancy between respondents in intervention and control groups at baseline, at 2 weeks and 6 weeks after educational intervention.
3. To compare TPB construct on adherence to daily iron intake between respondents in intervention and control groups at baseline, 2 weeks and 6 weeks after educational intervention.
4. To compare haemoglobin levels between respondents from intervention and control groups at baseline, 2 weeks and 6 weeks after educational intervention.
5. To compare dietary iron, vitamin C and caffeine intake between respondents from intervention and control group at baseline, 2 weeks and 4 weeks after educational intervention.

Design:

The study design will be a cluster randomized controlled trial. This study design was chosen as to avoid contamination of information between respondents from intervention and control groups that possible to occur if randomization of study subjects from the same antenatal clinic is conducted. Therefore, clusters i.e. antenatal clinics will be randomly assigned as intervention group and control group using randomization generator.

Setting:

Two antenatal clinics in Petaling district will be randomly selected as the study sites for this intervention study. One antenatal clinic will be randomly selected as intervention and another clinic will be control. Total duration of respondents' participation will be 6 weeks. Study population will be pregnant women who attend the selected antenatal clinics in Petaling district and have been diagnosed as anaemia. Sampling method will be multistage cluster sampling.

Inclusion criteria:

1. Age 20-40 years old
2. Women with pregnancy at 13-28 weeks gestation
3. Women diagnosed with anaemia with haemoglobin 7.0-10.9g/dl
4. Able to read and write in Malay and/or English
5. Participants have a smartphone installed with WhatsApp application

Exclusion criteria:

1. Symptomatic anaemia (breathlessness, chest pain, syncope, signs of heart failure)
2. Anemia due to thalassemia or other hematological disease
3. Anemia due to other diseases such as renal failure or cancer
4. Planned for termination of pregnancy

Respondents from intervention and control groups are matched for age (20 - 40 years old), gestational week (13 - 28 weeks of gestation) and haemoglobin level (7.0-10.9g/dL).

Intervention:

The intervention group will receive the "MyPinkMom" educational intervention which will be delivered through WhatsApp application as well as the routine antenatal care including iron supplement such as zincofer, maltofer, ferrous, iberet, or obimin. On the other hand, the control group will receive information on anaemia in pregnancy in antenatal card and same routine antenatal care as what intervention group received. The control group only received information on anaemia in pregnancy which is placed in the antenatal card.

The intervention will be carried out for 6 weeks. "MyPinkMom" educational intervention will be held at week 1. In each session, a respective "MyPinkMom" video with audio explanation will be delivered to respondents in intervention group through WhatsApp application. It will be delivered to respondents daily for 6 days and each video will take about 3-5 minutes duration. Sessions of "MyPinkMom" will cover general information on anaemia, pathophysiology of anaemia in pregnancy, proper nutrition, iron supplement therapy, possible side effect and how to overcome it as well as complications of anaemia on mothers and offspring.

Weekly reminder on proper dietary and iron supplement intake will be given trough WhatsApp at week 2 till week 5. Post-intervention assessment will be held at week 6.

Blinding:

Respondents and investigators will aware the intervention received by respondents. The data analysers will be blinded as they would not know respondents belongs to intervention or control group as each respondent will be labelled as numbers.

Evaluation of intervention Baseline test will be done before the intervention. Haemoglobin level at recruitment, sociodemographic, obstetric profile, dietary iron intake, knowledge score on anaemia in pregnancy, TPB construct on adherence to daily iron tablet intake will be determined at baseline.

Post-intervention test will be conducted at week 6. Haemoglobin level, knowledge score on anaemia in pregnancy, TPB construct on adherence to daily iron tablet intake, dietary iron, vitamin C and caffeine intake will be reassessed as post-intervention test. The haemoglobin level will be traced from the antenatal cards or from laboratory of respective clinics.

Outcomes of study

Primary outcomes:

Changes of haemoglobin level

Secondary outcomes:

1. Changes of knowledge score on anaemia in pregnancy score
2. Changes of Theory of Planned Behavior construct on adherence to daily iron tablet score changes
3. Changes of dietary iron, vitamin C and caffeine intake changes

Sample size calculation:

The sample size is calculated using the following formula for clinical trial:

n = 2(Zα+Z1-β)2σ2/Δ2 This gives the sample size per arm in a controlled clinical trial (n). In the formula, σ is estimated standard deviation and Δ is estimated effect size i.e. difference in effect noted between intervention and control group. For this study, the accepted p-value is less than 0.05 and study power is 80%. In this case, two-tailed test will be used as the results could be bidirectional. Therefore, value of Zα is 1.96 and Z1-β is 0.8416.

From previous study, the standard deviation would be approximately 0.8. From the same study, haemoglobin level increment in intervention group was 62.7% and in control group was 16.8%. The difference of haemoglobin level increment between intervention and control group were used to calculate the effect size (Δ). Thus, the effect size would be 45.9% (i.e., 0.459). The sample size for this study will be:

n = [2(1.96+0.8416)2(0.8)2] / (0.459)2 n=48 per arm Total sample size is 120 including 20% drop out (60 in intervention and 60 in control group).

Data analysis plan:

All categorical data will be analysed descriptively as frequency and percentage. All numerical data will be analysed as mean and standard deviation if normally distributed or as median and interquartile range if not normally distributed.

For baseline test, haemoglobin level, knowledge score on anaemia in pregnancy, TPB construct on adherence to daily iron tablet intake, dietary iron, Vitamin C and caffeine intake among participants from intervention and control group will be compared using Student t-test.

Comparison of haemoglobin level, knowledge score on anaemia in pregnancy, TPB construct on adherence to daily iron tablet, dietary iron, vitamin C and caffeine intake between intervention and control group at baseline and at week 6 will using paired t-test. Possible confounder will be controlled by conducting Multivariate ANOVA (MANOVA). Analysis will follow Intention to Treat analysis. Level of significance is at p-value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-40 years old
2. Women with pregnancy at 13-28 weeks gestation
3. Women diagnosed with anaemia with haemoglobin 7.0-10.9g/dl
4. Able to read and write in Malay and/or English
5. Participants have a smartphone installed with WhatsApp application

Exclusion Criteria:

1. Symptomatic anaemia (breathlessness, chest pain, syncope, signs of heart failure)
2. Anaemia due to thalassemia or other haematological disease
3. Anaemia due to other diseases such as renal failure or cancer
4. Planned for termination of pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women diagnosed with anaemia
Enrollment: 120 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
haemoglobin level changes | From baseline to week 8 (6 weeks post intervention)
  Haemoglobin level will be measure at baseline, at week 4 (2 weeks post intervention) and at week 8 (6 weeks post intervention). Change from baseline haemoglobin level at week 8 (6 weeks post intervention) between intervention and control groups will be evaluated. Haemoglobin level will be traced from full blood count result from respondents' antenatal cards or laboratory. Blood for full blood count is taken by trained staff respective clinics for every monthly antenatal visit.

SECONDARY OUTCOMES:
knowledge score changes | From baseline to week 8 (6 weeks post intervention)
  Knowledge level on anaemia in pregnancy will be evaluated at baseline, at week 4 (2 weeks post intervention) and at week 8 (6 weeks post intervention), using validated questionnaire of knowledge on anaemia in pregnancy. It contains 16 items. The items are statement related to anaemia in pregnancy. Responses for each item are 'True','False','Not sure'. 1 mark will be only given to correct answer. Incorrect answer and 'Not sure' answer will not be given marks. Total marks will be converted to percentage. Marks of 60-100 will be considered as good knowledge and marks of less than 60 will considered as poor knowledge. Change from baseline knowledge on anaemia in pregnancy at week 8 (6 weeks post intervention) between study groups will be evaluated.
Amount of dietary iron changes | From baseline to week 8 (6 weeks post intervention)
  Dietary iron intake will be measured at baseline, at week 4 (2 weeks post intervention) and at week 8 (6 weeks post intervention). This will be assessed using validated Pregnancy Food Frequency Questionnaire (FFQ). Amount of iron from diet will be presented in grams. Change from baseline amount of iron intake from diet at week 8 (6 weeks post intervention) between study groups will be determined.
Theory of Planned Behavior construct score changes | From baseline to week 8 (6 weeks post intervention)
  Theory of Planned Behavior construct score will be measured at baseline, at week 4 (2 weeks post intervention) and at week 8 (6 weeks post intervention). The score will be evaluated using validated Theory of Planned Behavior construct questionnaire. It contains 4 domains (intention, attitudes towards adherence to daily iron tablet, subjective norms and perceived behavior). It contains 17 items. Response for each item will be seven-point bipolar scale (1 to 7). '1' is 'strongly disagree' and '7' is 'strongly agree'. Change of Theory of Planned Behavior construct score on adherence to daily iron tablet intake from baseline to week 8 (6 weeks post intervention) between study groups will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Raudah Abd Rahman, MPH, Principal Investigator — Dr

IPD SHARING:
Plan to Share IPD: No